CLINICAL TRIAL: NCT04932278
Title: The Role of Osteopathic Manipulative Medicine in Recovery From Concussions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michigan State University (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Jacek Cholewicki, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY4542
Record Dates: First submitted 2021-06-11; First posted 2021-06-21 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Concussion, Brain
Keywords: concussion; Sport-related; Osteopathic manipulative treatment
MeSH Terms: conditions — Brain Concussion | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: For this study, participants will be randomly assigned to 1. Usual care, or 2. Usual care and OMT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Participants in this group will receive routine care for the management and treatment of concussions
  Interventions: Procedure: Usual care
- OMT Group (Experimental): Participants who are randomized into the OMT group will receive OMT in addition to their usual care.
  Interventions: Procedure: Osteopathic manipulative treatment; Procedure: Usual care

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment — Osteopathic manipulative treatment (OMT) is hands-on care provided by an osteopathic physician (D.O.). During osteopathic manipulative treatment, an osteopathic physician may move participants' muscles and joints using osteopathic techniques including stretching, gentle pressure and resistance, as well as thrust techniques that apply a quick, therapeutic force of brief duration that travels a short distance.
  Arms: OMT Group
Procedure: Usual care — Routine concussion management with healthcare professionals.

SUMMARY:
This project aims to study whether adding osteopathic manipulative treatment (OMT) to usual care of concussed patients will enhance their recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13-55 years
* Concussion sustained within the last 12 days

Exclusion Criteria:

* Contraindications to OMT, such as skull fracture, cervical fracture, signs of intracranial bleeding, or stroke
* Neck surgery within the last 6 months
* Any conditions recognized by a physician as contraindicating or impeding protocol implementation
* Will not be under the care of a healthcare professional
* Any active (or pending) worker's compensation, disability, or personal injury claims related to their concussion injury

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
SCAT5 symptom evaluation score | through study completion, up to 4 weeks
  Symptom evaluation score is a self-reported measure of the participants' post-concussion symptoms. Participants are scored on Total Number of Symptoms (ranges 0 to 22) and Symptom Severity Score (ranges 0 to 132). Higher scores represent worse outcome.

SECONDARY OUTCOMES:
Head position tracking accuracy | 2 weeks from injury
  Participants will be seated in an upright position with their upper body secured to a backrest and will wear a head harness with an attached position sensor. The angular position of the head will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by moving their head. Accuracy will be determined by taking the difference between the target position signal and the actual head position.
Head force tracking accuracy | 2 weeks from injury
  Participants will be seated in an upright position with their upper body secured to a backrest and will be asked to generate force with their head against a fixed pad. The pad will be attached to a load cell that monitors how much force is being generated by their head. The force level will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by generating force with their head. Accuracy will be determined by taking the difference between target force signal and the actual head force.
Return to play duration | through study completion, up to 4 weeks
  Number of days between injury date and receiving clearance to return to play or referred out to other specialists

CONTACTS AND LOCATIONS:
Locations (1):
- MSU Center for Orthopedic Research, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No